CLINICAL TRIAL: NCT02916810
Title: Alternative Stimulation Mode and Location for Auditory Hallucination Neuromodulation Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Xiaoming Du, Assistant Professsor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-24-0336; R61MH128390 (NIH)
Record Dates: First submitted 2016-06-28; First posted 2016-09-27 (Estimated); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia and Related Disorders
Keywords: transcranial magnetic stimulation; schizophrenia; MRI
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active rTMS stimulation (Active Comparator)
  Interventions: Device: Active rTMS stimulation
- Sham rTMS stimulation (Sham Comparator)
  Interventions: Device: Sham rTMS stimulation

INTERVENTIONS:
Device: Active rTMS stimulation — Participants will receive two rTMS sessions in each treatment visit for up to 22 visits within about 6 weeks. There is a 30-minute rest between the two rTMS sessions.
  Arms: Active rTMS stimulation
Device: Sham rTMS stimulation — Participants will receive two sham rTMS sessions in each treatment visit for up to 22 visits within about 6 weeks. There is a 30-minute rest between the two sham rTMS sessions.
  Arms: Sham rTMS stimulation

SUMMARY:
The purpose of the study is to test the hypothesis that functionally navigated repetitive TMS stimulations to the prefrontal cortex (PFC) modulate aberrant cortical electrical activities at PFC circuitry. The TMS location of the PFC site will be individually localized by the symptom-related functional connectivity between PFC and symptom related areas (such as the auditory and language processing cortex). The investigators predict that such modulation will correct abnormal activities in patients with schizophrenia, reduce symptoms, especially auditory hallucination, and improve working memory/sustained attention performance.

DETAILED DESCRIPTION:
Neuroimaging studies suggest that aberrant activities at specific brain regions such as sensory areas and language-related areas are related to psychosis symptoms including auditory and visual hallucination, delusion, and thought disorders. Transcranial magnetic stimulation (TMS) provides a non-invasive means for altering brain electrical neural activity. TMS has been approved by FDA for treatment of depression. Other applications have not been approved but it has been used in a wide range of clinical research especially in neurology and psychiatry. Among psychotic symptoms, there are preliminary significant improvement in treatments of auditory hallucination using TMS with small samples, but those treatments are not robust in larger samples. The high inter-subject variability limits the efficacy of TMS treatment in schizophrenia patients. The investigators aim to develop a TMS treatment method with a fMRI-defined treatment target area, where the TMS target is individually identified to maximize the TMS effects. The identification method uses both the anatomical character and its functional relationship with auditory hallucination and other psychosis symptoms. If the current target-identification successfully identified effective TMS target individually, the treatment efficacy will be significant improved and more patients will benefit from TMS treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ages between ages 18-50 years
* Ability to give written informed consent (age 18 or above)
* Diagnosed with schizophrenia-spectrum disorder and Evaluation to Sign Consent (ESC) above 10.
* Is currently under the care of a licensed primary care provider or mental healthcare provider (e.g., psychiatrist, psychologist, nurse practitioner, licensed clinical social worker).
* Have auditory hallucinations despite treated by two or more antipsychotics including one atypical antipsychotic medication.
* Agrees to: (a) provide written permission, as requested, to allow any and all forms of communication between the investigators and study staff and any health care provider who currently provides and/or has provided service to the subject within two years of study enrollment; and (b) provide the names and verifiable contact information (name, email and mailing address, mobile and land-line phone number, as applicable) of at least two reliable persons ≥ age 22, who reside within a 30-minute drive of the subject's residence, and whom the research staff is at liberty to contact, as deemed necessary, for the duration of study participation.

Exclusion Criteria:

* Persons with a first-degree relative with inherited epilepsy, seizure disorder, or seizures or persons who answer "yes" to any of the parts (A. - G.) of Question 3 of an epilepsy screening questionnaire.
* Taking > 400 mg clozapine/day and not on anti-seizure medication(s) with sufficient dose.
* Failed TMS screening questionnaire.
* Significant alcohol or other drug use (substance abuse within 1 month or substance dependence history within 6 months and having substance usage within 1 month) other than nicotine or marijuana dependence
* Any major medical illnesses that may affect normal brain functioning. Examples of these conditions include, but not limited to, stroke, CNS infection or tumor, other significant brain neurological conditions.
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* History of head injury with loss of consciousness over 10 minutes; history of brain surgery
* Cannot refrain from using alcohol and/or marijuana 24 hours or more prior to experiments.
* Woman who is pregnant (child-bearing potential but not on contraceptive and missing menstrual period; or by self-report; or by positive pregnancy test) or has had unprotected sexual intercourse without birth control in the last 4 weeks.
* Moderate-High Risk of suicide according to the Columbia - Suicide Severity Rating Scale (C-SSRS) Screen Version - Recent (i.e. answers YES to Question 3 and NO to Question 6 (Moderate risk); or answers YES to Questions 4, 5, or 6 (High risk) or in the clinical judgement of the investigator or the study psychiatrist.
* In the medical opinion of the investigator, subjects with the following circumstances or conditions which can increase the risk of seizures may be excluded: sleep deprivation; major depressive disorder comorbid with dementia, underweight status; concurrent use of cephalosporins and antiarrhythmics (particularly propranolol); metabolic abnormalities (hyponatremia, hypocalcemia, hypomagnesemia, hypoglycemia, hyperglycemia, renal failure/uremia, liver failure); raised blood concentrations of proconvulsant medications due to reduced clearance (e.g. secondary to initiation of antibiotics for treatment of infections); alcohol withdrawal; use of stimulants, such as cocaine or MDMA; use of immunosuppressive therapy with cyclosporine, tacrolimus and other agents that can cause the posterior reversible leukoencephalopathy syndrome; dialysis; systemic infection, and fever itself.
* History (or family history) of deep vein thrombosis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Brain connectivity as indicated by resting state functional connectivity value as assessed by functional magnetic resonance imaging (fMRI) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  Functional magnetic resonance imaging (fMRI) is used to evaluate the brain activities that are corresponding to the treatment effect on auditory hallucination.

SECONDARY OUTCOMES:
Electrophysiological responses as indicated by mismatch negativity amplitudes from electroencephalography recording (EEG) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  Electroencephalogram (EEG) is used to evaluate the brain electrical activities that are corresponding to the treatment effect on auditory hallucination.
Electrophysiological responses as indicated by steady-state auditory evoked potentials from electroencephalography recording (EEG) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  Electroencephalogram (EEG) is used to evaluate the brain electrical activities that are corresponding to the treatment effect on auditory hallucination.
Auditory hallucinations as assessed by Psychotic Symptom Rating Scale (PSYRATS) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  Total score ranges from 0 to 44, with a lower score indicating a better outcome.
Negative symptoms as assessed by Brief Negative Symptom Scale (BNSS) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  Total score ranges from 0 to 90, with a lower score indicating a better outcome.
Cognitive insight as assessed by the Beck Cognitive Insight Scale (BCIS) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  Total score ranges from 15 to 60, with a lower score indicating a better outcome.
Depression as assessed by the Beck Depression Inventory measures the severity of depression | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  Total score ranges from 0 to 63, with a lower score indicating a better outcome.
Depression as assessed by the Calgary Depression Scale for Schizophrenia (CDSS) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  Total score ranges from 0 to 27, with a lower score indicating a better outcome.
Perception as assessed by the Perception State and Trait Scales (State score) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  The Perception State and Trait Scale measures subtle auditory and visual anomalies. State total score ranges from 0 to 48, with a lower score indicating a better outcome.
Perception as assessed by the Perception State and Trait Scales (Trait score) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  The Perception State and Trait Scale measures subtle auditory and visual anomalies. Trait total score ranges from 0 to 48, with a lower score indicating a better outcome.
Delusion as assessed by the Peters Delusions Inventory (yes/no score) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  The Peters Delusions Inventory measures subtle delusional tendencies. Yes/No total score ranges from 0 to 21, with a lower score indicating a better outcome.
Delusion as assessed by the Peters Delusions Inventory (distress score) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  The Peters Delusions Inventory measures subtle delusional tendencies. Distress total score ranges from 0 to 105, with a lower score indicating a better outcome.
Delusion as assessed by the Peters Delusions Inventory (pre-occupation score) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  The Peters Delusions Inventory measures subtle delusional tendencies. Pre-occupation total score ranges from 0 to 105, with a lower score indicating a better outcome.
Delusion as assessed by the Peters Delusions Inventory (conviction score) | baseline, intermittent (before or at the beginning of treatment visit 11, about 2 weeks after baseline), end of acute treatment (after treatment visit 20, about 4 weeks after baseline)
  The Peters Delusions Inventory measures subtle delusional tendencies. Conviction total score ranges from 0 to 105, with a lower score indicating a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Du, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No